CLINICAL TRIAL: NCT05363800
Title: Phase I Study of HRS-3738 in Recurrent and Refractory Non-Hodgkin's Lymphoma and Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-3738-I-102
Record Dates: First submitted 2022-04-25; First posted 2022-05-06 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-04

CONDITIONS: Recurrent and Refractory Non-Hodgkin's Lymphoma and Multiple Myeloma
MeSH Terms: conditions — Recurrence; Lymphoma, Non-Hodgkin; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Single arm study of HRS-3738
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-3738 (Experimental): In dose Escalation:
  HRS-3738 will be taken in oral. Seven dose levels are preset.
  In dose Expansion:
  2 to 3 dose cohorts will be selected for dose expansion stage.
  In indication Expansion:
  Indications will be selected to evaluate preliminary efficacy.
  Interventions: Drug: HRS-3738

INTERVENTIONS:
Drug: HRS-3738 — HRS-3738 will be administrated per dose level in which the patients are assigned.

SUMMARY:
This study is an open-label, multicenter Phase I clinical trial to evaluate the safety, tolerability, pharmacokinetics and efficacy of HRS-3738 in patients with recurrent and refractory Non-Hodgkin's lymphoma and multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Active multiple myeloma in accordance with IMWG criteria，or histopathologically and immunohistochemically confirmed non-Hodgkin's lymphoma in accordance with the 2016 WHO Classification of lymphoid neoplasias.
2. Recurred or did not alleviate after the previous treatment.
3. Have at least one measurable lesion.
4. With a life expectancy of ≥3 months.
5. Male or female ≥ 18 years old.
6. ECOG performance status of 0-1.
7. Subjects must voluntarily agree to participate in the trial and sign a written informed consent form.

Exclusion Criteria:

1. Amyloidosis, plasma cell leukemia.
2. Corrected serum calcium>3.4mmol/L(13.5mg/dl).
3. Presence of metastasis to central nervous system.
4. Treatment of other investigational products.
5. Major surgical therapy within 28 days prior to the date of signature of informed consent form, or expected major surgery during the study.
6. Known history of hypersensitivity to any components of HRS-3738.
7. Other factors that may affect the study results or lead to forced termination of the study early as judged by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | From Day 1 to Day 28
  Incidence and category of dose limiting toxicities (DLTs) during the first 28-day cycle of HRS-3738 treatment.
RP2D | From Day 1 to Day 28
  RP2D will be determined on the basis of evaluation on safety, PK, efficacy data in dose escalation and dose expansion stages.

SECONDARY OUTCOMES:
Safety endpoints: adverse events(AEs), serious adverse events（SAEs） | From Day 1 to 30 days after last dose.
  Assess safety and tolerability of HRS-3738 by way of adverse events (CTCAE v5.0).
Efficacy endpoints: Overall response rate (ORR) | From Day 1 to 30 days after last dose.
  Evaluated using Lugano 2014 criteria and IMWG criteria.
Efficacy endpoints: Best of response (BOR) | From Day 1 to 30 days after last dose
  Evaluated using Lugano 2014 criteria and IMWG criteria
Efficacy endpoints: time to response (TTR) | From Day 1 to 30 days after last dose.
  Evaluated using Lugano 2014 criteria and IMWG criteria.
Efficacy endpoints: Duration of response (DoR) | From Day 1 to 30 days after last dose
  Evaluated using Lugano 2014 criteria and IMWG criteria
Efficacy endpoints: Progression-free survival (PFS) | From Day 1 to 30 days after last dose
  Evaluated using Lugano 2014 criteria and IMWG criteria
Efficacy endpoints: overall survival (OS). | From Day 1 to 30 days after last dose.
  Evaluated using Lugano 2014 criteria and IMWG criteria.
Cmax | From Day 1 to 30 days after last dose
  Maximal plasma concentration
Tmax | From Day 1 to 30 days after last dose
  Time to Cmax
AUC | From Day 1 to 30 days after last dose
  Area under the plasma concentration-time curve
t1/2 | From Day 1 to 30 days after last dose
  Terminal-phase elimination half-life
Vz/F | From Day 1 to 30 days after last dose
  Apparent volume of distribution during terminal phase after non-intravenous administration
CL/F | From Day 1 to 30 days after last dose
  Apparent total clearance of the drug from plasma after oral administration.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Henan cancer Hospital, Zhengzhou, Henan
  - Sheng Jing Hospital of China Medical University, Shengyang, Liaoning
  - Zhejiang University School of Medicine The First Affiliated Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided